CLINICAL TRIAL: NCT02279537
Title: A Retrospective and Prospective Non-interventional Open Label Study to Assess the Real Life of Treatment-naive Patients With Wet Age-related Macular Degeneration in Routine Clinical Practice in France and Starting an Anti VEGF Therapy With Aflibercept
Brief Title: Real Life of Aflibercept In FraNce: oBservatiOnnal Study in Wet AMD
Acronym: RAINBOW
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 17374; EY1411FR (Other: Company Internal)
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Wet Macular Degeneration
Keywords: Wet age-related macular Degeneration (Wet-AMD); Naïve patients; Real life; Aflibercept
MeSH Terms: conditions — Wet Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: According to the recommendations of the Summary of Product Characteristics (SmPC)
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Administration by intravitreal injection

SUMMARY:
The purpose of this study is to collect real-life data on patients with wet age related macular degeneration (AMD) for whom treatment with Eylea was initiated

DETAILED DESCRIPTION:
The study is both retrospective and prospective to collect local real life data on patients under routine treatment. The observation period starts on January 2014. Patients who have received the 1st injection with Eylea from January 2014 will be enrolled.

Patients will be followed up for a period of 48 months or until it is no longer possible

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of wet AMD will be enrolled after the decision for treatment with Aflibercept (Eylea) has been made
* Patient with 1st injection of Eylea from 01 January 2014 until 30 April 2015 will be enrolled
* Prior/current treatment with any anti-VEGF intravitreal injections or macular laser (laser and/or visudyne/PDT) in the fellow eye is allowed
* Man or woman aged 18 years or more
* Patient who has been given appropriate information about the study objectives and procedures and who has given his/her written, informed consent;

Exclusion Criteria:

* Patient with another retinal disease: diabetic retinopathy, diabetic macular oedema (DME), myopic choroidal neovascularization, retinal vein occlusion (RVO), central serous chorioretinopathy (CSC), angioid streaks
* Patient who does not meet the local indication criteria for Eylea treatment.Contraindications listed in the Summary of Product Characteristics (SmPC) must be taken into account
* Patient who has previously been treated with any macular laser (laser and/or visudyne/PDT) or any anti-VEGF intravitreal injections for the study eye
* Patient taking part in an interventional study at the time of enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Naïve treatment patients with wet AMD who started a treatment with Anti VEGF (Vascular Endothelial Growth Factor) may be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 593 (Actual)
Dates: Start 2014-01-02 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Change in the measurement of best-corrected visual acuity (BCVA) from baseline to 12 months. | Baseline to 12 months
  As assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) method or any visual logarithmic scale

SECONDARY OUTCOMES:
Change in Best Corrected Visual Acuity (BCVA) during the second year and until the fourth year of treatment versus the initial visit | Baseline to 2 year, 3 year, 4 year
Percentage of patients who experienced a gain in BCVA, from initial visit to each follow-up visit (letter score of ≥ 0 letters, ≥ 5 letters, ≥ 10 letters, ≥ 15 letters) | Baseline to 1 year, 2 year, 3 year, 4 year
Percentage of patients losing fewer than 15 letters from the initial visit visual acuity at each follow-up visit | Baseline to 1 year, 2 year, 3 year, 4 year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, France

REFERENCES:
- [Result] Cohen SY, Dominguez M, Coscas F, Faure C, Baillif S, Oubraham H, Kodjikian L, Weber M; RAINBOW study investigators. Final 4-year results of the RAINBOW real-world study: intravitreal aflibercept dosing regimens in France in treatment-naive patients with neovascular age-related macular degeneration. Graefes Arch Clin Exp Ophthalmol. 2023 Apr;261(4):959-969. doi: 10.1007/s00417-022-05900-6. Epub 2022 Nov 18. PMID 36399178
- [Derived] Weber M, Kodjikian L, Coscas F, Faure C, Aubry I, Dufour I, Cohen SY. Impact of intravitreal aflibercept dosing regimens in treatment-naive patients with neovascular age-related macular degeneration in routine clinical practice in France: results from the RAINBOW study. BMJ Open Ophthalmol. 2020 Apr 6;5(1):e000377. doi: 10.1136/bmjophth-2019-000377. eCollection 2020. PMID 32518833
- [Derived] Weber M, Dominguez M, Coscas F, Faure C, Baillif S, Kodjikian L, Cohen SY. Impact of intravitreal aflibercept dosing regimens in treatment-naive patients with neovascular age-related macular degeneration: 2-year results of RAINBOW. BMC Ophthalmol. 2020 May 25;20(1):206. doi: 10.1186/s12886-020-01468-z. PMID 32450838
- [Derived] Weber M, Velasque L, Coscas F, Faure C, Aubry I, Cohen SY; RAINBOW study investigators. Effectiveness and safety of intravitreal aflibercept in patients with wet age-related macular degeneration treated in routine clinical practices across France: 12-month outcomes of the RAINBOW study. BMJ Open Ophthalmol. 2019 Apr 9;4(1):e000109. doi: 10.1136/bmjophth-2017-000109. eCollection 2019. PMID 31179386